CLINICAL TRIAL: NCT00231647
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Parallel-Group Study to Assess the Efficacy and Safety of Topiramate OROS Controlled-Release in the Treatment of Obese, Type 2 Diabetic Subjects Managed With Diet or Metformin
Brief Title: A Study on Efficacy and Safety of Topiramate OROS Controlled-Release in Obese, Type 2 Diabetic Subjects Managed With Diet or Metformin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002674
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-01

CONDITIONS: Obesity; Diabetes Mellitus, Type 2; Diabetes Mellitus, Adult-Onset
Keywords: Obesity; Type 2 Diabetes Mellitus; Metformin; Diabetic Diet; Topiramate; Adult-Onset Diabetes Mellitus (AODM)
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of a topiramate controlled-release formulation in the treatment of obese, type 2 diabetic patients managed with diet alone or combined with metformin.

DETAILED DESCRIPTION:
Topiramate is not approved for the treatment of obesity. Studies have shown that an immediate release formulation of topiramate reduces body weight in obese patients with or without type 2 diabetes. A novel controlled-release formulation of topiramate using OROS® technology has the potential for better efficacy and safety in the treatment of obesity. This double-blind, placebo controlled study will evaluate the effectiveness and safety of the controlled-release formulation in the treatment of obese subjects with type 2 diabetes. The study consists of 2 screening visits, a baseline visit, 7-week titration phase (topiramate dose will be increased from 25mg daily to 175mg daily), 9-week maintenance phase, 2-week taper phase and a 2-week follow-up. Effectiveness will be evaluated by the percent change in body weight, body mass index, and anthropometric measurements (waist and hip circumferences and their ratio). Safety evaluations (incidence and severity of adverse events, physical measurements and clinical laboratory tests) will be conducted throughout the study. The study hypothesis is that topiramate 175 mg daily, when administered as the OROS® controlled-release formulation, is effective (in terms of percent reduction in body weight from baseline to week 16) and safe, as compared with placebo, in the treatment of obese, type 2 diabetic patients managed with either diet alone or combined with metformin. During the titration phase, topiramate (in the OROS® controlled-release formulation) will be gradually increased to 175mg daily by mouth, and the dose will be maintained for 9 weeks, and then slowly discontinued over 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) >= 27 kg/m^2 and <50 kg/m^2
* Diagnosis of type 2 diabetes, managed with either diet alone or combined with monotherapy treatment with metformin
* Stable weight for at least 2 months
* Female patients must be postmenopausal for at least 1 year, surgically incapable of childbearing, practicing abstinence, or practicing an acceptable method of contraception (requires negative pregnancy test).

Exclusion Criteria:

* Contraindication or hypersensitivity to topiramate
* Exposure to any other experimental drug or device within past 90 days
* Established diagnosis of Type 1 diabetes
* History of severe or recurrent hypoglycemic episodes prior to study entry
* Taking oral antidiabetic medications other than metformin
* Treatment with insulin within 4 months
* Significant liver, kidney or cardiovascular diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2004-02; Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Percent change in body weight from baseline to Week 16.

SECONDARY OUTCOMES:
Changes in body weight, body mass index,anthropometric measurements (waste and hip circumference and their ratio),fasting blood glucose and lipid profile from baseline to Week 16; safety evaluations including incidence of adverse events during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Study on Efficacy and Safety of Topiramate OROS� Controlled-Release in Obese Type 2, Diabetic Subjects Managed with Diet or Metformin — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=486&filename=CR002674_CSR.pdf